CLINICAL TRIAL: NCT02765321
Title: Populational Program of Physical Activity and Healthy Eating Promotion: the "Life of Health" Study
Acronym: Life of Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Life of Health Study
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical activity and healthy eating promotion (Experimental)
  Interventions: Behavioral: Healthy lifestyle promotion

INTERVENTIONS:
Behavioral: Healthy lifestyle promotion — Healthy lifestyle changes (i.e., increase in physical activity levels and improvement in eating habits) will be promoted via population-based counselling through media (i.e., radio, newspapers, magazines, television, banners), cell phone applicative, workshops, specific programs at schools and companies, and community physical activity programs.

SUMMARY:
This is a population-based "natural experiment" study aimed to examine the effect of a multi-approach intervention focused on physical activity and healthy eating promotion to individuals living in Jaguariuna city (São Paulo, Brazil).

ELIGIBILITY:
Inclusion Criteria:

* citizens from Jaguariuna city (Sao Paulo, Brazil)

Exclusion Criteria:

* citizens not from Jaguariuna city (Sao Paulo, Brazil)
* children below 8 years of age.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
waist circumference | 7 months

SECONDARY OUTCOMES:
fasting glycemia | 7 months
fasting insulinemia | 7 months
total cholesterol | 7 months
LDL-cholesterol | 7 months
HDL-cholesterol | 7 months
triglycerides | 7 months
VLDL-cholesterol | 7 months
C-reactive protein | 7 months
objectively measured physical activity levels | 7 months
  assessed by accelerometers in a sub-sample
subjectively measured physical activity levels | 7 months
  assessed by International Physical Activity Questionnaires (IPAQ)
subjectively measured physical activity levels | 7 months
  assessed by phone interview
food intake | 7 months
  food frequency questionnaire
blood pressure | 7 months
body mass index | 7 months
self-perceived health status | 7 months
  assessed by phone interview

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana B Benatti, PhD, Principal Investigator — University of Sao Paulo; Marcio Atalla, Principal Investigator — Casa do BemStar Marcio Atalla; Evelyn F Costa, PhD, Principal Investigator — University of Sao Paulo; Alex Florindo, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No